CLINICAL TRIAL: NCT00745472
Title: The Amplitude of Auditory Evoked Potentials and the Intensity of Experimental Pain Stimulation in Healthy Volunteers
Brief Title: Auditory Evoked Potentials and Experimental Pain
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Thomas P. Enggaard MD, PHD, Department of Anaesthesiology, Odense University Hospital, Denmark
Other Study IDs: 30071993
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Pain
Keywords: AEP; experimental pain; healthy volunteers
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Monitoring of auditory evoked potentials (AEP) in patients during general anaesthesia is commonly used to ensure a sufficient hypnotic level during surgery. The amplitude of AEP (AEPa) has in clinical settings been found to correlate to pain. The aim of the study was to test, if AEPa could detect increasing experimental pain stimulations in healthy volunteers. Electric nerve stimulation, cold and heat pain were used as pain models.

DETAILED DESCRIPTION:
During the AEP monitoring, healthy volunteers were exposed to experimental pain. At study day 1: Firstly, single electric nerve stimulation and repetitive electric nerve stimulations causing temporal pain summation. The stimulations were given at 50, 75 and 100% of the thresholds for pain tolerance and temporal pain summation. Secondly, the volunteers were exposed to cold pain by use of two different Cold Pressor Tests (CPT) with water temperatures at 8 and 1 Celsius. All measurements were repeated after an hour to test reproducibility.

At study day 2: Brief Thermal Stimulation were used with two different temperatures and duration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 20 - 40 years old

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
VAS and amplitude of AEP | before, during and after experimental pain

SECONDARY OUTCOMES:
reproducibility | after an hour

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Enggaard, MD, Principal Investigator — Odense University Hospital